CLINICAL TRIAL: NCT02829827
Title: An Open-label Adaptive Study for the Assessment of Safety, Tolerability, Pharmacokinetics, and Efficacy of Multiple Doses of Radiprodil in Subjects With Drug-resistant Infantile Spasms
Brief Title: A Phase 2 Study of Radiprodil in Subjects With Drug-resistant Infantile Spasms (IS)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: After reviewing the feasibility and projected completion date of the study, UCB has made the decision to stop the study
Sponsor: UCB Biopharma S.P.R.L. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EP0078; 2016-002107-26 (EudraCT Number)
Record Dates: First submitted 2016-07-08; First posted 2016-07-12 (Estimated); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Infantile Spasms (IS)
Keywords: Radiprodil; Infantile spasms; IS; Infantile; Spasms; Epilepsy; Paediatrics; Drug-resistant; West Syndrome; Hypsarrhythmia
MeSH Terms: conditions — Spasms, Infantile; Spasm; Epilepsy | interventions — radiprodil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiprodil (Experimental): Each subject will enter an individualized dose titration schedule.
  Interventions: Drug: Radiprodil

INTERVENTIONS:
Drug: Radiprodil — Radiprodil at individualized doses.

SUMMARY:
The purpose of the study is to evaluate the safety and tolerability, the pharmacokinetics and the efficacy of radiprodil in abolishing clinical spasms in subjects with drug-resistant infantile spasms

DETAILED DESCRIPTION:
The study is divided into 3 parts:

Part A - exploratory, Part B - confirmatory, Part C - open label extension

ELIGIBILITY:
Inclusion Criteria:

Part A and B:

* Subject is male or female between 2 and 14 months of age
* The diagnosis of infantile spasms (IS)
* Subject has drug-resistant IS

Part C:

* Subject participated in EP0078 Part A and received 2 radiprodil treatment cycles
* Subject experienced a relapse of spasms during the down taper or within 5 half-lives (3 days) discontinuation of radiprodil treatment in Cycle 2 of Part A
* Electroencephalogram (EEG) on baseline Part C is compatible with the diagnosis of infantile spasms

Exclusion Criteria:

Part A and B:

* More than 6 months have passed since the diagnosis of Infantile Spasms (IS)
* Current treatment with cannabinoids
* Subject has hematocrit greater than 60
* Subject has any medical condition that, in the opinion of the Investigator, could jeopardize or would compromise the subject's ability to participate in this study
* Subject has a history or current condition predisposing to respiratory dysfunction
* Current treatment with felbamate
* Current treatment with perampanel
* Ketogenic diet
* Clinically significant lab abnormalities
* Clinically significant abnormality on ECG that, in the opinion of the Investigator, increases the safety risks of participating in the study
* Subject has a lethal or potentially lethal condition other than IS, with a significant risk of death before 18 months of age such as non-ketotic hyperglycinemia
* Body weight is below 4 kg
* Known history of severe anaphylactic reaction secondary to medication intake or serious blood dyscrasias

Part C:

* Subject experienced any acute tolerability issues in either treatment cycle in Part A which the investigator and the sponsor medical monitor consider a risk for further participation
* Subject met any withdrawal criteria in Part A
* Subject has experienced any adverse effects or developed any new medical conditions since enrollment in Part A which the investigator considers could significantly increase the safety risks of participating in Part C

Ages: 2 Months to 14 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2018-10-02 (Actual); Study Completion 2018-10-02 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with clinical response on Day 14 of treatment with the maintenance dose of radiprodil | Day 14, counting from the first day of radiprodil at maintenance dose
  Clinical response is defined as no spasms on Day 14 of treatment with the maintenance dose of radiprodil. This is the primary efficacy variable for Part A.
Estimates of exposure generated from a population-Pharmacokinetic modelling | Samples will be taken at baseline (time during Day -14 to -1 prior to dosing) and 3, 4, 5 & 12hr after the 1st dose on Day 1 of radiprodil low, mid & high dose. Blood samples will be taken at same timepoints after 1st dose on Day 2 of radiprodil low dose
  This is a primary variable for Part A.
Percentage of subjects with electro-clinical response on Day 14 of treatment with the maintenance dose of radiprodil | Day 14, counting from the first day of radiprodil at maintenance dose
  Electro-clinical response is defined as no spasms and resolution of hypsarrythmia on Day 14 of treatment with the maintenance dose of radiprodil. This is the primary efficacy variable for Part B.
Incidence of Adverse Events (AEs) during the study | From Baseline (Day -1) to the end of the Post-treatment Period (28 days post last dosing)
  An AE is any untoward medical occurrence in a subject or trial subject that is administered a drug or biologic (medicinal product) or that is using a medical device. The event does not necessarily have a causal relationship with that treatment or usage. This is a primary variable for all parts.

SECONDARY OUTCOMES:
Percentage of subjects with electro-clinical response on Day 14 of treatment with the maintenance dose of radiprodil | Day 14, counting from the first day of radiprodil at maintenance dose
  Electro-clinical response is defined as no spasms and resolution of hypsarrythmia on Day 14 of treatment with the maintenance dose of radiprodil. This is the secondary efficacy variable for Part A.
Percentage of subjects with clinical response on Day 14 of treatment with the maintenance dose of radiprodil | Day 14, counting from Day 14 of treatment with the maintenance dose of radiprodil
  Clinical response is defined as no spasms on Day 14 of treatment with the maintenance dose of radiprodil. This is the secondary efficacy variable for Part B.
Estimates of exposure generated from a population-Pharmacokinetic modelling | Pharmacokinetic samples will be collected on Day 1 of radiprodil low dose, mid dose and high dose. Additionally, blood samples will be taken after 1st dose on Day 2 of radiprodil low dose.
  This is a secondary variable for Part B.
Time to cessation of spasms | During the first 14 days of treatment with radiprodil
  Time to cessation of spasms for clinical responders on Day 14 of treatment with the maintenance dose of radiprodol. This is a secondary efficacy variable for parts A and B.
Percentage of responders with clinical relapse | 12 months, counting from Day 14 of treatment with the maintenance dose of radiprodil
  The percentage of clinical responders on Day 14 of treatment with the maintenance dose of radiprodil with clinical relapse within 12 months. This is a secondary efficacy variable for parts A and B.
Time to clinical relapse from the day of spasm cessation | From day of spasms cessation up to 42 months of age
  This is a secondary efficacy variable for parts A and B.
Percentage of electro-clinical responders with electro-clinical relapse | 12 months, counting from Day 14 of treatment with the maintenance dose of radiprodil
  The percentage of electro-clinical responders on Day 14 of treatment with the maintenance dose of radiprodil with electro-clinical relapse within 12 months. This is a secondary efficacy variable for parts A and B.
Time to electro-clinical relapse from the day of spasm cessation | From day of spasms cessation up to 42 months of age
  This is a secondary efficacy variable for parts A and B.
Percentage of subjects with extended clinical response | 28 days, counting from Day 14 (inclusive) of treatment with the maintenance dose of radiprodil
  Extended clinical response is defined as no spasms for 28 consecutive days from Day 14 of treatment with the maintenance dose of radiprodil. This is a secondary efficacy variable for parts A and B.
Percentage of subjects with extended electro-clinical response | 28 days, counting from Day 14 (inclusive) of treatment with the maintenance dose of radiprodil
  Extended electro-clinical response is defined as no spasms and resolution of hypsarrythmia for 28 consecutive days from Day 14 of treatment with the maintenance dose of radiprodil. This is a secondary efficacy variable for parts A and B.
Percentage of subjects with extended clinical response to each additional treatment cycle on Day 14 of treatment with the maintenance dose of radiprodil | 28 days, counting from Day 14 (inclusive) of maintenance dose
  Extended clinical response is defined as no spasms for 28 consecutive days from Day 14 of treatment with the maintenance dose of radiprodil. This is a secondary efficacy variable for part C.
Number of treatment cycles per subject | During Part C (Day -1 to Day 28 of the Maintenance Period)
  This is a secondary variable for Part C.
Percentage of subjects with electro-clinical response to each additional treatment cycle on Day 14 of treatment with the maintenance dose of radiprodil | Day 14, counting from the first day of maintenance dose
  Electro-clinical response is defined as no spasms and resolution of hypsarrythmia on Day 14 of treatment with the maintenance dose of radiprodil. This is a secondary efficacy variable for Part C.
Time to clinical relapse from the first day of no witnessed spasms for each treatment cycle | From day of no witnessed spasms up to 42 months of age
  This is a secondary efficacy variable for part C.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — +1 8445992273 (UCB)
Locations (1):
- Ep0078 401, Paris, France